CLINICAL TRIAL: NCT03891407
Title: Acceptability and Feasibility of Unsupervised HIV Self-Testing Among Networks of Men:Tanzania STEP (Self-Testing Education and Promotion) Project
Brief Title: Acceptability and Feasibility of Unsupervised HIV Self-Testing Among Networks of Men
Acronym: STEP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of South Carolina (Other)
Responsible Party: Principal Investigator, Donaldson Conserve, PhD, Study Coordinator for Donaldson Conserve, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Pro00072005
Record Dates: First submitted 2019-02-26; First posted 2019-03-27 (Actual); Last update posted 2020-11-25 (Actual); Status verified 2020-11

CONDITIONS: HIV Infections; HIV/AIDS; Hiv
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Intervention Model Description: Participants who agree to self-test will receive pretest counseling and a 10 minute demonstration, including a video in addition to verbal instructions, of how to use an oral self-test kit from a trained HIV counselor. After counseling, participants will receive 2 oral fluid self-test kits to conduct the self-test at home or in a private location during the next 3 months, a phone number to call in case they need assistance when performing the self-test at home, and a location where to return the used self-test kits and collect more test kits throughout the study period. Upon returning the used self-test kits after every 3 months, participants will be able to share their self-test result with the counselor. Participants will also be asked at each pick-up time to demonstrate they can use the kit to ensure participants continue to receive correct self-test results throughout the study period.
Masking Description: Peer-led recruitment strategy.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- HIV Self-testing Group (Experimental): Camp members will receive information about HIV self-testing from peer educators who will be nominated by you and other camp members in your camp. Camp members in the STEP project will receive pretest counseling and a 10 minute demonstration. They will receive 1 oral fluid HIV self-test kit to conduct the self-test at home or in a private location during the next 1 month and a phone number to call in case you need assistance when performing the self-test at home. They will also receive information about the nearest HIV Care and Treatment Center where they can seek a confirmatory HIV test and start HIV treatment in the event of a positive self-test result.
  Interventions: Diagnostic Test: Self-Testing Education and Promotion
- Non-intervention Group (No Intervention): Camp members will be encouraged to seek HIV testing at the clinics.

INTERVENTIONS:
Diagnostic Test: Self-Testing Education and Promotion — Camp members will receive the Self-Testing Education and Promotion (STEP locally referred to as Mate Yako Afya Yako) intervention and will receive HIV-counseling and oral HIV self-testing kits.
  Arms: HIV Self-testing Group

SUMMARY:
The purpose of this study is to recruit and train men to promote HIV self-testing to their network members in their camps and examine the efficacy of a peer-led HIV self-testing intervention on the uptake of HIV testing among men.

DETAILED DESCRIPTION:
The research is the first evaluation of an unsupervised HIV self-testing strategy in Tanzania focusing on networks of heterosexual men. The reasons for focusing on heterosexual men is because heterosexual contact is the primary mode of HIV transmission in Tanzania and data from our previous trial indicate that 97% of the male camp members are heterosexual. Moreover it will be the first intervention to engage male peer leaders to promote HIV self-testing in their social networks in Tanzania. We will build on previous work our research team has conducted to identify 'camps' or local venues where young men socialize with elected leaders and members pay membership dues. Our previous intervention has proven successful to recruit and train leaders from camps to serve as community health leaders in their respective camps, with the goal of changing social norms related to HIV and gender-based violence. A novel approach to the proposed research is that we will leverage the work we have conducted within camps with social networks of men to test the acceptability and feasibility of oral fluid-based HIV self-testing and confirmatory blood-based HIV testing within existing networks of men that we know we can access through stable social venues. We will recruit male camp leaders to train them about HIV self-testing and instruct them to return to their camps and engage their male peers by informing them about HIV self-testing for prior to our research team offering participants the opportunity to self-test.

ELIGIBILITY:
Inclusion Criteria:

* Participant is at least 18 years old
* Has been member of the camp for at least 3 months
* Visits camp at least once a week
* Intends to live in Dar es Salaam for next 6 months
* Has not had suicidal thoughts in the past
* Willing to give contact information of self and relative or friend

Exclusion Criteria:

* Does not meet all inclusion criteria
* Unable to participate due to psychological disturbance, cognitive impairment or threatening behavior

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male members of participating camps.
Enrollment: 500 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
Number of HIV self-testing kits distributed in the past 3 Months | 3 months
  Camp members' use of the HIV self-testing kits will be evaluated at 3 months

SECONDARY OUTCOMES:
Number of camp members who self-report HIV self-testing in the past 3 months | 3 months
  Camp members will self-report HIV self-testing at 3 Months

CONTACTS AND LOCATIONS:
Locations (1):
- Tandale Community, Dar es Salaam, Tanzania